CLINICAL TRIAL: NCT03829605
Title: Plasma Measurement of Hydrogen Sulfide, Nitric Oxide and Stress Hyperglycemia in Acute Myocardial Infarction
Brief Title: Plasma Hydrogen Sulfide, Nitric Oxide and Stress Hyperglycemia in Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham I El-mahdy, Principal Investigator, Assiut University
Other Study IDs: Myocardial infarction
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Myocardial Infarction
Keywords: Hydrogen sulfide; Nitric oxide; Stress hyperglycemia; Acute coronary syndrome
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I:: Fifty AMI patients on admission
  Interventions: Other: Measurement of hydrogen sulfide
- Group II:: The previous AMI patients after 12 hours
  Interventions: Other: Measurement of hydrogen sulfide

INTERVENTIONS:
Other: Measurement of hydrogen sulfide — Hydrogen sulfide will be measured by ELISA and correlated with nitric oxide and hyperglycemia

SUMMARY:
Acute myocardial infarction (AMI) can cause heart failure, an irregular heartbeat, cardiogenic shock, or cardiac arrest. It is the major cause of morbidity and mortality in the general population. The diagnosis of AMI is complex basing on the clinical history, physical examination, cardiac markers, and a chest radiograph. Besides, considering that the mechanisms linking activation of inflammation and ACS are complex as well, progress in diagnosis and therapy improves little

DETAILED DESCRIPTION:
The World Health Organization (WHO) indexed cardiovascular disease (CVD) as a leading foundation for human death in developing as well as developed countries. Ischemic necrosis of the myocardium is called myocar¬dial infarction. Despite improvements in medical and interventional therapies in recent years, acute myocar¬dial infarction is still an important cause of mortal¬ity and morbidity. Hydrogen sulfide (H2S) is a colorless, water-soluble gas and is an endogenously produced labile diffusible mediator with multiple roles in the cardiovascular system in health and disease. H2S is endogenously generated, and cystathionine-β-synthase (CBS), cystathionine-γ-lyase (CSE), and 3-mercaptopyruvate sulfurtransferase (3-MST) are key enzymes involved in its biological production. Once interacting with carbon monoxide and nitric oxide, H2S will initiate a unique gaseous signaling net¬work and participate in the regulation of multiple patho¬physiological processes. Plasma H2S levels negatively correlated with HbA1c, duration of diabetes, and systolic and diastolic blood pressures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of AMI-
* Patients of age 18 years or more who are willing to participate in the study and give their consent for same.

Exclusion Criteria:

* Patients with congenital heart diseases, alcoholics with a past history of liver disease, pulmonary embolus, sepsis, chest trauma, and renal failure were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Acute myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2019-04-20 (Estimated); Study Completion 2019-05-20 (Estimated)

PRIMARY OUTCOMES:
The mean difference of hydrogen sulfide before and after treatment | 12 hours
  Hydrogen sulfide mean difference will be measured by ELISA in myocardial infarction.

REFERENCES:
- [Background] Suzuki K, Sagara M, Aoki C, Tanaka S, Aso Y. Clinical Implication of Plasma Hydrogen Sulfide Levels in Japanese Patients with Type 2 Diabetes. Intern Med. 2017;56(1):17-21. doi: 10.2169/internalmedicine.56.7403. Epub 2017 Jan 1. PMID 28049995
- [Background] Peter EA, Shen X, Shah SH, Pardue S, Glawe JD, Zhang WW, Reddy P, Akkus NI, Varma J, Kevil CG. Plasma free H2S levels are elevated in patients with cardiovascular disease. J Am Heart Assoc. 2013 Oct 23;2(5):e000387. doi: 10.1161/JAHA.113.000387. PMID 24152982
- [Background] Kuang Q, Xue N, Chen J, Shen Z, Cui X, Fang Y, Ding X. Low Plasma Hydrogen Sulfide Is Associated with Impaired Renal Function and Cardiac Dysfunction. Am J Nephrol. 2018;47(5):361-371. doi: 10.1159/000489606. Epub 2018 May 18. PMID 29779029
- [Background] Marfella R, Siniscalchi M, Esposito K, Sellitto A, De Fanis U, Romano C, Portoghese M, Siciliano S, Nappo F, Sasso FC, Mininni N, Cacciapuoti F, Lucivero G, Giunta R, Verza M, Giugliano D. Effects of stress hyperglycemia on acute myocardial infarction: role of inflammatory immune process in functional cardiac outcome. Diabetes Care. 2003 Nov;26(11):3129-35. doi: 10.2337/diacare.26.11.3129. PMID 14578250